CLINICAL TRIAL: NCT00004656
Title: Nutritional Aspects of Rett Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Baylor College of Medicine (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Diagnostic
Other Study IDs: 199/11814; BCM-CNRC-H1637
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-02

CONDITIONS: Rett Syndrome
Keywords: Rett syndrome; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Rett Syndrome; Neurologic Manifestations; Mental Disorders; Rare Diseases

INTERVENTIONS:
Procedure: Metabolic assessment with body composition evaluation

SUMMARY:
OBJECTIVES: I. Determine dietary macronutrient intake in children with Rett syndrome and in healthy controls.

II. Measure sleeping and awake metabolic rates in various positions, i.e., reclining, sitting, and standing, by whole-room indirect calorimetry and isotope dilution.

III. Quantify activity patterns by time-motion studies using 24-hour activity records and 12-hour videotaping.

IV. Correlate 24-hour activity patterns with 24-hour heart rate telemetry and short-term oxygen consumption.

V. Estimate 24-hour fecal and urinary energy losses. VI. Determine body composition by clinical anthropometry, whole-body potassium counting, and total-body electrical conductance.

VII. Calculate apparent energy needs based on measurement of energy intake and expenditure.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

All participants undergo extensive nutritional and metabolic assessment with body composition evaluation. Studies include macronutrient intake, body fat, lean muscle mass, metabolic rate, and time-action studies; and 24-hour cardiac telemetry. Rett syndrome girls also receive a hemogram and hand x-ray.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

Patients aged 5 to 18 with Rett syndrome Able to sleep and awaken alone

Ages: 5 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Dates: Start 1993-05

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen J. Motil, Study Chair — Baylor College of Medicine